CLINICAL TRIAL: NCT05450588
Title: Development and Validation of Waist Girth Based-equations to Evaluate Body Composition in Colombian Population With Different Physical Activity Levels - F20 Project
Brief Title: Development and Validation of Equations to Evaluate Body Composition in Colombian Population - F20 Project
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dynamical Business and Science Society - DBSS International SAS (Network)
Collaborators: CES University (Other); Universidad de Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: Acta0031Proy115TG; DBSS_F20_CES (Other: DBSS International SAS)
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Body Composition; Obesity
Keywords: Body composition; Waist Girth; Regression Ecuations; Fat mass; Fat free mass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sedentary: It will be obtained by open call for both students and administrative staff at the CES University.
- Physically active: Under the collaboration framework bet ween DBSS international SAS and Smart Fit Colombia, a sample of personal trainers who reside and work in Medellín, or its metropolitan area will be invited to participate.
- Athletes: Under the collaboration framework between DBSS international SAS and ARTHROS Physiotherapy and Exercise Center, a sample of professional athletes from different sports disciplines will be invited to participate.

SUMMARY:
The assessment of body composition is one of the main components within the evaluation of nutritional status under the ABCDE model. Generally, the use of equations to estimate components is a frequent strategy since it represents a doubly indirect method that has good correlation with methods of higher sensitivity (i.e., NMR, DXA, etc.). In this sense, the waist girth or circumference (WC) represents a quick, simple and inexpensive tool to evaluate the excess of fat mass in the human being; however, this measurement does not provide information on body composition in isolation and has been used as an important independent variable in some recent equations (e.g., relative fat mass [RFM]). Considering the lack of formulas or external validation of RFM in the Colombian population, the aim of this STROBE-Nut-based cross-sectional study is to develop and validate simple equations that use WC as an independent variable to estimate fat mass and fat-free mass in a population with different physical activity levels.

DETAILED DESCRIPTION:
This research aims to validate and develop WC-based equations due to the estimation potential to assess body composition in the athletic, physically active and sedentary Colombian population. We will follow the standardized reporting guidelines of the Strengthening the Reporting of Observational Studies in Epidemiology-Nutritional Epidemiology (STROBE-nut). Stratified probability sampling techniques will be used. Participants of >18 years old, residing in Medellín or its metropolitan area, with different physical activity levels, and that give consent to be evaluated by health professionals will be invited to participate. Anthropometry and DXA assessment will be carried out in the participants. Subsequently, validation of the RFM will be performed by comparing the estimation results with gold standard methods using correlation and agreement (Bland-Altman) analyses. Finally, several models will be developed to estimate fat mass and fat-free mass in the population subgroups (athletes, physically active individuals and sedentary people). The results of this research will improve professional practice in health, exercise and sports science.

The F20 project is developed by the Research Division of the Dynamical Business & Science Society-DBSS International SAS with the support of University CES, University de Córdoba, University Distrital Francisco José de Caldas, Exercise & Sport Nutrition Laboratory at Texas A&M University, the R&D department of ARTHROS IPS, Smart Fit, and IPS Diagnosticarte.

ELIGIBILITY:
Inclusion Criteria:

1. +18 years old (under 60 years)
2. Sedentary, Physically active and Athletes of competitive level.
3. Residing in the city of Medellín or nearby municipalities of the metropolitan area.
4. Signed informed consent.
5. Assist to anthropometric and DXA measurements.

Exclusion Criteria:

1. People with a disease and/or special condition that limits exposure to radiation emitted by DXA.
2. Adults over 60 years of age
3. Pregnant women
4. Athletes with injuries
5. People with implants or prostheses.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: According to previous recommendations (Knofczynski and Mundfrom,2007), 130 participants will be needed to obtain a coefficient of determination (R2) of 0.5 with an excellent level of prediction and with three independent variables. The subjects will be divided into three groups for validation and development of the new equations, the total number of participants will be divided into 3 strata following optimal allocation methods. Assigned a fixed cost for each stratum (sedentary people, C1; physically active subjects, C2; and sportsmen, C3, given that C3>C2>C1).The values obtained for the sedentary group were n=54, the physically active population group n= 43, and the sportsmen group n=33. In the new equation, the development/validation ratio will be 70/30 over the number of subjects.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Two-component model of body composition (fat mass and free mass) | One year (March 2024 to June 2024)
  Through DXA measurement and the estimation using anthropometry-based equations.

SECONDARY OUTCOMES:
Anthropometry-based morphological | One year (March 2024 to June 2024)
  Analysis to compare Colombian population with different physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Bonilla, PhD, Principal Investigator — Research Division, DBSS International SAS.; Jorge L Petro, PhD, Study Chair — Research Division, DBSS International SAS.; Laura P Muñoz, MSc, Study Director — Grupo de Investigación Nutral, Facultad Ciencias de la Nutrición y los Alimentos, Universidad CES.; Leidy T Duque, MSc, Study Director — Grupo de Investigación Nutral, Facultad Ciencias de la Nutrición y los Alimentos, Universidad CES.
Locations (1):
- Ces Nutral, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonilla DA, Duque-Zuluaga LT, Munoz-Urrego LP, Moreno Y, Velez-Gutierrez JM, Franco-Hoyos K, Agudelo-Martinez A, Humeres G, Kreider RB, Petro JL. Development and Validation of Waist Girth-Based Equations to Evaluate Body Composition in Colombian Adults: Rationale and STROBE-Nut-Based Protocol of the F20 Project. Int J Environ Res Public Health. 2022 Aug 27;19(17):10690. doi: 10.3390/ijerph191710690. PMID 36078407
- See also: Defining cutoffs to diagnose obesity using the relative fat mass (RFM): Association with mortality in NHANES 1999-2014 — https://pubmed.ncbi.nlm.nih.gov/31911664/
- See also: Body shape indices are predictors for estimating fat-free mass in male athletes — http://pubmed.ncbi.nlm.nih.gov/31649287/